CLINICAL TRIAL: NCT04971239
Title: The Efficacy and Safety of Topical Methotrexate Microemulsion in Combination With Excimer Light and Narrow Band-ultraviolet B in the Treatment of Plaque Psoriasis
Brief Title: Topical Methotrexate Microemulsion in the Treatment of Plaque Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Mahmoud Abdelsalam, Ayat Mahmoud Abdel Salam, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTXPSORIASIS
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis; Methotrexate
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- topical methotrexate microemulsion (Active Comparator): Group(A): topical methotrexate micro emulsion formulation, each patient will be instructed to apply a very thin film of 0.5 ml of it over the three psoriatic plaques three times weekly .
  Interventions: Drug: topical methotrexate micoemulsion
- combination of topical methotrexate microemulsion and excimer light (Experimental): Group(B) : excimer laser will be done twice weekly on a different psoriatic plaques in combination with topical methotrexate micro emulsion for a total treatment course of 12 weeks.
  Interventions: Drug: topical methotrexate micoemulsion; Device: Excimer light
- combination of topical methotrexate microemulsion and narrow band-ultraviolet B (Experimental): Group(C) : Narrow band ultraviolet B will be done twice weekly on a different psoriatic plaques in combination with topical methotrexate micro emulsion for a total treatment course of 12 weeks
  Interventions: Drug: topical methotrexate micoemulsion; Device: Narrow band ultraviolet B

INTERVENTIONS:
Drug: topical methotrexate micoemulsion — The selected microemulsion composition consists of 40% Jojoba oil, 45% Tween-80 and Span-85 at a ratio of 3:1 as surfactant and co surfactant, respectively and 15% water. The chosen concentration was based on preliminary studies conducted which delineated that these ratios provided the best skin deposition based on factorial skin modelling.The prepared microemulsions contains 0.1% methotrexate
  Other Names: Methotrexate nano-emulsion
Device: Excimer light — the excimer laser will be done twice weekly for a total treatment course of 12 weeks.
  Arms: combination of topical methotrexate microemulsion and excimer light
Device: Narrow band ultraviolet B — the Narrow band ultraviolet B will be done twice weekly for a total treatment course of 12 weeks.
  Other Names: NB-UVB
  Arms: combination of topical methotrexate microemulsion and narrow band-ultraviolet B

SUMMARY:
* Psoriasis is a chronic relapsing dermatological disease which often necessitates a long-term therapy and occurs in a significant percent of the population . It affects the skin and sometimes the nails and joints of patients .
* Psoriatic patients are frequently categorized into two groups: mild or moderate to severe psoriasis, depending on the clinical severity of the lesions, the percentage of affected body surface area, and patient quality of life .
* Topical drug therapy is the cornerstone in the treatment of mild to moderate psoriasis. It offers a direct targeting of affected skin by avoiding systemic adverse events .
* Several topical therapies are available for the treatment of psoriasis such as topical steroid , topical vitamin D3 analogues (calcipotriol),tar, anthraline, topical tacrolimus (a non-steroidal calcineurin inhibitor) and tazarotene (a third-generation retinoid) . However, they do not provide an adequate response owing to the inadequate percutaneous absorption and poor patient compliance caused by greasiness and stickiness of some formulations, and some patients even remain untreated .
* So that, patient satisfaction with available topical treatments remains modest .

DETAILED DESCRIPTION:
* Methotrexate was US Food and Drug Administration approved for the treatment of psoriasis, and is currently recommended for practically all forms of moderate or severe psoriasis, including psoriatic arthritis .
* Methotrexate competitively inhibits dihydrofolate reductase enzyme which converts dihydrofolate to tetrahydrofolate (fully reduced folic acid); the latter being a necessary cofactor in the synthesis of DNA . Because systemic Methotrexate is associated with several adverse effects, topical Methotrexate has become a more-interesting alternative .
* However, the topical action of Methotrexate is challenging, since it suffers limited percutaneous diffusivity owing to its aqueous solubility, its ionization at physiological pH, and unfavorable lipid/water coefficient .
* A remedy to this problem might be the utilization of a suitable customized nano-based delivery system for enhancing the topical percutaneous penetration of MTX for treatment of psoriasis .
* Micro emulsions are among the most promising nanocarriers, being composed of aqueous and oily phases in addition to surfactants and cosurfactants . Only one study used micro emulsion as a topical nanocarrier for MTX, and jojoba oil will be selected as the oily phase of the micro emulsion since it exhibits moisturizing and anti-inflammatory effects which are beneficial in psoriasis treatment .
* The physical therapies used for the treatment of psoriasis include PUVA, broad band ultraviolet ray, Narrowband ultraviolet B and monochromatic excimer laser and light.
* Narrowband ultraviolet B (307-311 nm) showed efficacy in the treatment of psoriasis. This therapeutic approach considers that psoriasis patients undergoing phototherapy usually receive high cumulative doses of radiation during their lives, thus leading to secondary cutaneous disorders, like photoaging, telangiectasias, excessive tanning .
* On the contrary, The monochromatic excimer light device delivers ultraviolet B wavelength at 308 nm only to the lesional skin, could lower all these collateral effects dramatically and decreasing the total dose of radiation. Moreover, the treatment may be tailored to each affected area with different doses of ultraviolet makes monochromatic excimer laser and light mostly appreciated to a large part of patients, thus increasing treatment compliance, which is particularly useful when we have to deal with long-lasting therapeutic protocols.
* Finally, the possibility to focus the radiations on skin lesions is believed to reduces the risks of acute and chronic side effects in the uninvolved safe skin
* Several studies showed its effectiveness in the treatment of psoriasis as a monotherapy or in combination with several topical therapies such as flumetasone, dithranol, calcipotriol , but no study investigate its efficacy in combination with topical methotrexate yet.
* In recent years, the new biological therapies (monoclonal antibodies, receptor fusion proteins and similar) have been developed to manage psoriasis in its inner mechanisms of immune regulation. However, the legal (i.e. FDA and EMA-approved use of biologics in psoriasis) and scientific limitations (i.e. guidelines) for the use of biologics, together with the major possible medical involvements connected to this category of therapeutic agents and their expensive cost, make of them a treatment dedicated to a few well-chosen patients .

ELIGIBILITY:
Inclusion criteria:

1. Thirty patients with mild psoriasis will be recruited from the Dermatology Outpatient Clinic, Assiut University Hospital.
2. The diagnosis will be based upon the clinical characteristics of plaque psoriasis.
3. Patients will be included after they have stopped any systemic therapy for at least 8 weeks and topical therapy for at least 2 weeks.

Exclusion Criteria:

1. Patients having cardiovascular, renal or liver diseases.
2. Patients with photosensitive or psychological disorders or immunodeficient patients.
3. Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
percentage of clinically improved patients using psoriasis severity index | three months
  clinical assessment using psoriasis severity index

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Goff KL, Karimkhani C, Boyers LN, Weinstock MA, Lott JP, Hay RJ, Coffeng LE, Norton SA, Naldi L, Dunnick C, Armstrong AW, Dellavalle RP. The global burden of psoriatic skin disease. Br J Dermatol. 2015 Jun;172(6):1665-1668. doi: 10.1111/bjd.13715. Epub 2015 May 6. No abstract available. PMID 25645671
- [Result] Mrowietz U, Kragballe K, Reich K, Spuls P, Griffiths CE, Nast A, Franke J, Antoniou C, Arenberger P, Balieva F, Bylaite M, Correia O, Dauden E, Gisondi P, Iversen L, Kemeny L, Lahfa M, Nijsten T, Rantanen T, Reich A, Rosenbach T, Segaert S, Smith C, Talme T, Volc-Platzer B, Yawalkar N. Definition of treatment goals for moderate to severe psoriasis: a European consensus. Arch Dermatol Res. 2011 Jan;303(1):1-10. doi: 10.1007/s00403-010-1080-1. Epub 2010 Sep 21. PMID 20857129
- [Result] Wollina U, Tirant M, Vojvodic A, Lotti T. Treatment of Psoriasis: Novel Approaches to Topical Delivery. Open Access Maced J Med Sci. 2019 Aug 30;7(18):3018-3025. doi: 10.3889/oamjms.2019.414. eCollection 2019 Sep 30. PMID 31850114
- [Result] Abdelgawad R, Nasr M, Moftah NH, Hamza MY. Phospholipid membrane tubulation using ceramide doping "Cerosomes": Characterization and clinical application in psoriasis treatment. Eur J Pharm Sci. 2017 Apr 1;101:258-268. doi: 10.1016/j.ejps.2017.02.030. Epub 2017 Feb 21. PMID 28232140
- [Result] Florek AG, Wang CJ, Armstrong AW. Treatment preferences and treatment satisfaction among psoriasis patients: a systematic review. Arch Dermatol Res. 2018 May;310(4):271-319. doi: 10.1007/s00403-018-1808-x. Epub 2018 Feb 13. PMID 29442137
- [Result] Carretero G, Puig L, Dehesa L, Carrascosa JM, Ribera M, Sanchez-Regana M, Dauden E, Vidal D, Alsina M, Munoz-Santos C, Lopez-Estebaranz JL, Notario J, Ferrandiz C, Vanaclocha F, Garcia-Bustinduy M, Taberner R, Belinchon I, Sanchez-Carazo J, Moreno JC; Grupo de Psoriasis de la AEDV. [Guidelines on the use of methotrexate in psoriasis]. Actas Dermosifiliogr. 2010 Sep;101(7):600-13. Spanish. PMID 20858386
- [Result] Ramez SA, Soliman MM, Fadel M, Nour El-Deen F, Nasr M, Youness ER, Aboel-Fadl DM. Novel methotrexate soft nanocarrier/fractional erbium YAG laser combination for clinical treatment of plaque psoriasis. Artif Cells Nanomed Biotechnol. 2018;46(sup1):996-1002. doi: 10.1080/21691401.2018.1440236. Epub 2018 Feb 15. PMID 29448838
- [Result] Ali MF, Salah M, Rafea M, Saleh N. Liposomal methotrexate hydrogel for treatment of localized psoriasis: preparation, characterization and laser targeting. Med Sci Monit. 2008 Dec;14(12):PI66-74. PMID 19043379
- [Result] Wong TW, Zhao YL, Sen A, Hui SW. Pilot study of topical delivery of methotrexate by electroporation. Br J Dermatol. 2005 Mar;152(3):524-30. doi: 10.1111/j.1365-2133.2005.06455.x. PMID 15787822
- [Result] Nasr M, Abdel-Hamid S, Moftah NH, Fadel M, Alyoussef AA. Jojoba Oil Soft Colloidal Nanocarrier of a Synthetic Retinoid: Preparation, Characterization and Clinical Efficacy in Psoriatic Patients. Curr Drug Deliv. 2017;14(3):426-432. doi: 10.2174/1567201813666160513132321. PMID 27174314
- [Result] Gianfaldoni S, Gianfaldoni R, Wollina U, Lotti J, Tchernev G, Lotti T. An Overview on Radiotherapy: From Its History to Its Current Applications in Dermatology. Open Access Maced J Med Sci. 2017 Jul 18;5(4):521-525. doi: 10.3889/oamjms.2017.122. eCollection 2017 Jul 25. PMID 28785349
- [Result] Mehraban S, Feily A. 308nm excimer laser in dermatology. J Lasers Med Sci. 2014 Winter;5(1):8-12. PMID 25606333
- [Result] Langley RG, Ellis CN. Evaluating psoriasis with Psoriasis Area and Severity Index, Psoriasis Global Assessment, and Lattice System Physician's Global Assessment. J Am Acad Dermatol. 2004 Oct;51(4):563-9. doi: 10.1016/j.jaad.2004.04.012. PMID 15389191